CLINICAL TRIAL: NCT04912960
Title: Application of PEEP in Patients With Acute Respiratory Failure Caused by Lung Injury: Assessment of Clinical Practice
Brief Title: PEEP in Patients With Acute Respiratory Failure
Status: Recruiting | Type: Observational
Sponsor: Jesus Villar (Other)
Responsible Party: Sponsor-Investigator, Jesus Villar, Principal investigator, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: 170090
Record Dates: First submitted 2021-05-24; First posted 2021-06-03 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Acute Respiratory Failure With Hypoxia
MeSH Terms: interventions — Respiration, Artificial; Positive-Pressure Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mechanical ventilation — Optimum PEEP
  Other Names: positive end-expiratory pressure

SUMMARY:
Positive end-expiratory pressure (PEEP) has become an essential component of the care of critically ill patients who require ventilatory support. In 1975, several investigators published the effects of PEEP in 15 mechanically ventilated patients with acute respiratory failure (ARF) supported by mechanical ventilation. FiO2 ranged between 21% to 75% and the tidal volume between 13 to 15 mL/kg. PEEP was increased in 3 cmH2O steps until cardiac output fell. The aim was to identify the "optimum" PEEP level. "Best" PEEP was associated simultaneously with the best static compliance of the respiratory system, the greatest oxygen transport, and the lowest dead space fraction. That study established the basis for the use of PEEP in patients with ARF worldwide. Although currently patients with ARF are ventilated with much lower tidal volumes, that study has never been validated. It is unknow whether their findings are currently valid, generalizable, and reproducible.

DETAILED DESCRIPTION:
With the application of PEEP, the baseline end-expiratory pressure in mechanically ventilated patients is elevated above atmospheric pressure. PEEP is applied generally to improve oxygenation, which is usually not observed unless there is a concomitant increase in the functional residual capacity, probably by preventing airway closure and recruiting previously unventilated alveoli.

Fifty years later, we have improved our knowledge on lung physiology and pulmonary mechanics in patients requiring mechanical ventilation (MV). To date, most ARF patients on MV are managed with incremental PEEP levels.

The team of investigators in this study has postulated that it is appropriate to assess whether the routine clinical practice of applying increasing levels of PEEP pursues the best oxygenation and the best compliance, or by contrary, it was a random finding by investigators back in 1975. For the current assessment of this approach at the bedside (gradual increase of PEEP to identify the optimum level of PEEP), the investigators cannot reproduce exactly that approach since current recommendations for ventilating patients with severe ARF include: (i) the use of tidal volumes between 4-8 ml/kg predicted body weight, (ii) monitoring cardiac output using a pulmonary artery catheter is not a routine clinical practice in critically ill patients, and (iii) measuring dead space fraction is not part of the routine management of patients with acute respiratory failure.

The investigators in this study will assess in 15 mechanically ventilated patients with ARF whether the highest lung compliance during the identification of optimal PEEP in each patient coincides with the level of best oxygenation and ventilation. PEEP levels will be individualized in each patient, as part of common practice in the Post-Surgical Critical Care Unit of the hospital. Data from 15 patients requiring MV for >24 h due to ARF will be analyzed to identify the optimum PEEP level. Only data from patients in which the cause of ARF is of pulmonary origin (atelectasis, lung contusion, aspiration of gastric content, and lung infection) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Intubated patients requiring MV for >24 h
* Age >18 years
* Acute hypoxemic respiratory failure, defined as a PaO2/FiO2 <300 with an FiO2 ≥0.3 and PEEP≥5 cmH2O.
* ARF caused by pulmonary insults.

Exclusion Criteria:

* ARF from non-pulmonary origin.
* Contraindications from high PEEP (severe head trauma or severe chest trauma).
* Patients that cannot maintained supine position.
* Uncorrected hypovolemia
* Hemodynamic instability

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients with hypoxemic respiratory failure (PaO2/FiO2 <300 on FiO2 equal or greater than 0.3)
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
static compliance of the respiratory system | at study enrollment
  ratio of tidal volume to pressure gradiente of the respiratory system
oxygen transport | at study enrollment
  Cardiac output multiply by oxygen content in arterial blood
dead space fraction | at study enrollment
  ratio of dead space to tidal volume

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, MD, Study Director — Hospital Universitario Dr. Negrin
Locations (3):
- Spain (3):
  - Hospital Universitario Dr. Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Clinic, Barcelona
  - Hospital Universitario La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: No
data collection will be shared with all study investigators

REFERENCES:
- [Background] Suter PM, Fairley B, Isenberg MD. Optimum end-expiratory airway pressure in patients with acute pulmonary failure. N Engl J Med. 1975 Feb 6;292(6):284-9. doi: 10.1056/NEJM197502062920604. PMID 234174
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162